CLINICAL TRIAL: NCT00491387
Title: Sympathetic Nervous System Modulation in Hypertension by Beta-adrenergic Blockade
Brief Title: Sympathetic Nervous System Modulation in Hypertension
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Adverse events reported with beta-blockers as primary therapy.
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Myron C. Gerson, Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #07-01-12-01
Record Dates: First submitted 2007-06-21; First posted 2007-06-26 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Hypertension
Keywords: hypertension; sympathetic nervous system
MeSH Terms: conditions — Hypertension | interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- metoprolol succinate (Experimental): Subjects will undergo I-123 MIBG testing before and after sustained-release beta-adrenergic blockade.
  Interventions: Drug: Metoprolol Succinate

INTERVENTIONS:
Drug: Metoprolol Succinate — Once daily, oral, 12.5 mg to 200 mg, dose titrated to reduce heart rate by 20% or to less than 65 beats per minute.
  Other Names: Toprol XL; metoprolol XR

SUMMARY:
This is a study of patients with high blood pressure who are already treated with an angiotensin converting enzyme inhibitor or receptor blocker and have achieved good or fair blood pressure control. The hypothesis is that addition of the beta-adrenergic receptor blocker, sustained-release metoprolol, will provide additional blockade of the sympathetic nervous system, thereby further improving left ventricular filling and blood pressure control.

DETAILED DESCRIPTION:
Patients were to receive sympathetic cardiac innervation testing with I-123 MIBG at baseline and again after receiving a titrate dose of beta-blocker. Data were to be assesses by repeated measures testing.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension with blood pressure less than 140/90 on either an ACE inhibitor or angiotensin receptor blocker

Exclusion Criteria:

* Known valvular heart disease of more than mild severity
* Known coronary artery disease defined by an angiographic coronary artery stenosis greater than or equal to 50% luminal diameter narrowing, acute or previous myocardial infarction, or previous coronary revascularization
* Known non-ischemic cardiomyopathy with left ventricular ejection fraction less than 50%
* Atrial fibrillation
* Current treatment with a β-adrenergic blocking drug or a calcium channel blocker
* Current treatment with a psychoactive or other drug known to alter 123I-MIBG uptake
* Participation in another research study within the prior 30 days
* A life-limiting disease process that is likely to preclude completion of study participation
* Pregnancy or breast feeding
* Inability or unwillingness to provide informed consent
* Baseline resting heart rate less than 65 beats per minute
* Diabetes
* Iodine allergy
* Unwilling to sign informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron C Gerson, M.D., Principal Investigator — University of Cincinnati

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was stopped early due to concerns resulting from a publication reporting an increased in mortality in cardiac deaths in patients treated with beta-blockers as the primary drug for hypertension. Although no adverse reactions were observed in the present study, it was decided by the PI that beta-blockers could not ethically be continued.
Groups:
- Group 1: Treated with metoprolol succinate
Period: Overall Study
Arm/Group | Group 1
Started | 24
Study Enrollment | 24
Completed | 4
Not Completed | 20
Not completed — study terminated | 20

BASELINE CHARACTERISTICS:
Groups:
- Metoprolol Succinate: will receive I-123 MIBG innervation imaging before and after metoprolol succinate
Arm/Group | Metoprolol Succinate
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Sympathetic Cardiac Innervation as Measured by I-123 MIBG Heart - Mediastinum Ratio
Description: 24 subjects had baseline I-123 MIBG imaging. No subject completed all aspects of the protocol. The study was closed due to unfavorable publication related to metoprolol treatment for hypertension.
Time Frame: january 2018
Arm/Group | Metoprolol Succinate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Metoprolol Succinate: Patients receive I-123 MIBG imaging before and after metoprolol succinate.
Arm/Group | Metoprolol Succinate
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

LIMITATIONS AND CAVEATS:
Early termination due to a publication in the literature suggesting potential increased cardiac mortality in hypertensive patients treated primarily with beta blockers. Did not feel that continued treatment in volunteer subjects could be justified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No